CLINICAL TRIAL: NCT00959244
Title: 1) Effects of Therapeutic Agents on Estrogens in the Breast 2) Utilizing the Resources of the Breast Cancer Collaborative Registry (BCCR)
Brief Title: Study of Urine Samples From Women With Newly Diagnosed Breast Cancer Enrolled on Clinical Trial UNMC-08105
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0502-08-EP; P30CA036727 (NIH)
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Chromatography, High Pressure Liquid; Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: high performance liquid chromatography — Analyses of urine will be conducted by ultraperformance liquid chromatography with detection by tandem mass spectrometry.
Other: laboratory biomarker analysis — The biomarkers of interest will be the metabolites 4-OHE1(E2), estrogen-GSH conjugates and depurinating estrogen-DNA adducts.
Other: mass spectrometry — Analyses of urine will be conducted by ultraperformance liquid chromatography with detection by tandem mass spectrometry.
Other: medical chart review — Information about age, race, general health, any endocrine disorders, history of cancer, estrogen and progesterone receptor status, menopausal status and breast disease, body mass index, age at menarche, menopausal status (pre- or peri- menopausal or postmenopausal), age at menopause if applicable, chemotherapy regimen (if applicable), radiation therapy (if applicable), smoking history, alcohol consumption, pregnancy history including age at each pregnancy, lactation, history of benign breast disease, hysterectomy and disease type.

SUMMARY:
RATIONALE: Studying samples of urine from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at urine samples from women with newly diagnosed breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To learn the effects of selected agents (tamoxifen and aromatase inhibitors) on the profile of estrogen metabolites, glutathione conjugates, and depurinating DNA adducts in urine from women with breast cancer.

OUTLINE: Previously collected urine samples are analyzed for 40 estrogen metabolites, conjugates, and depurinating DNA adducts by ultra-performance liquid chromatography with tandem mass spectrometric detection.

Patient information (e.g., race, body mass index, age at menarche, menopausal status, age at menopause if applicable, smoking history, alcohol consumption) is collected through medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ductal carcinoma in situ or invasive breast cancer
* Urine biospecimens available from participation in protocol UNMC-08105 (IRB#311-06), the Breast Cancer Collaborative Registry (BCCR), which included treatment with tamoxifen or an aromatase inhibitor

  o Urine specimens were collected at baseline, 6 months, and then annually
* Estrogen receptor or progesterone receptor positive
* ECOG performance status 0-2

Exclusion Criteria:

* Not pregnant or nursing
* No concurrent use of estrogen(s)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-02-02 (Actual); Primary Completion 2009-09-25 (Actual); Study Completion 2009-09-25 (Actual)

PRIMARY OUTCOMES:
Estrogen compounds | at baseline at 6 months and annually
  Estrogen compounds in urine

CONTACTS AND LOCATIONS:
Overall Officials: Ercole Cavalieri, DSc, Principal Investigator — Eppley Cancer Center, University of Nebraska Medical Center
Locations (1):
- Eppley Cancer Center, University of Nebraska Medical Center, Omaha, Nebraska, United States